CLINICAL TRIAL: NCT02634073
Title: An Open-label Single-Center, 4-Period William's Cross-Over Design Drug Interaction Trial to Determine the Effects of Sorbitol-Containing Solutions on Lamivudine Exposure Following Administration of Lamivudine Oral Solution in Healthy Adult Subjects
Brief Title: A Phase IV, Open Label, 4-period Cross-over Study to Investigate a Drug Interaction Between Lamivudine and Sorbitol Oral Solutions in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 204857
Record Dates: First submitted 2015-12-14; First posted 2015-12-17 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-02

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: Lamivudine; Safety; Sorbitol; Pharmacokinetics
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — Lamivudine; Sorbitol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment A: Lamivudine 300 milligram(mg) (Experimental): Participant will receive single dose of Lamivudine 300 mg (30 ml of 10 mg/ml Oral Solution) after overnight fasting. Treatment period will be separated by at least 7 day wash out period.
  Interventions: Drug: Lamivudine
- Treatment B: Lamivudine 300 mg + Sorbitol 3.2 g (low dose) (Experimental): Participant will receive single dose of Lamivudine 300 mg (30 ml of 10 mg/ml Oral Solution) + oral solution of Sorbitol 3.2 g after overnight fasting. Treatment period will be separated by at least 7 day wash out period.
  Interventions: Drug: Lamivudine; Drug: Sorbitol
- Treatment C: Lamivudine 300 mg + Sorbitol 10.2 g (medium dose) (Experimental): Participant will receive single dose of Lamivudine 300 mg (30 ml of 10 mg/ml Oral Solution) + oral solution of Sorbitol 10.2 g after overnight fasting. Treatment period will be separated by at least 7 day wash out period
  Interventions: Drug: Lamivudine; Drug: Sorbitol
- Treatment D: Lamivudine 300 mg + Sorbitol 13.4 g (high dose) (Experimental): Participant will receive single dose of Lamivudine 300 mg (30 ml of 10 mg/ml Oral Solution) + oral solution of Sorbitol 13.4 g after overnight fasting. Treatment period will be separated by at least 7 day wash out period
  Interventions: Drug: Lamivudine; Drug: Sorbitol

INTERVENTIONS:
Drug: Lamivudine — It is a clear, colorless to pale yellow solution with the odour of fruit. It will be provided in a 240 mL bottle with the strength of 10 mg/mL Lamivudine 300 mg (30 mL of solution) will be administered orally to the participants
Drug: Sorbitol — It is a clear, colorless, odourless solution. It will be available in 3 dosage levels viz;. 3.2 g (low dose), 10.2 g (medium dose) and 13.4 g (high dose) sorbitol total dose.
  Arms: Treatment B: Lamivudine 300 mg + Sorbitol 3.2 g (low dose); Treatment C: Lamivudine 300 mg + Sorbitol 10.2 g (medium dose); Treatment D: Lamivudine 300 mg + Sorbitol 13.4 g (high dose)

SUMMARY:
Lamivudine (3TC) is a nucleoside analogue indicated in combination with other antiretroviral agents for the treatment of human immunodeficiency virus type 1 (HIV-1) infection in adults and children. Documented literature elucidates that simultaneous administration of multiple sorbitol-containing products could increase the potential for a significant interaction and may contribute to the lower 3TC exposures.

In this study several sorbitol doses (3.2 gram (g), 10.2 g, and 13.4 g solutions) will be administered with lamivudine to investigate dose dependency and mimic the situation where multiple sorbitol-containing antiretroviral medications may be co-administered with lamivudine. It will be open label, randomized, 4-way crossover (by William's design method) design at a single centre. Randomized participants will receive a single dose of each of four treatments after wash out period of minimum 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age inclusive, at the time of signing the informed consent.
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination and laboratory tests.
* A participant with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator in consultation with the Medical Monitor if required agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight >=50 kilogram (kg) (110 pounds [lb]) for men and >45 kg (99 lb) for women and body mass index (BMI) within the range 18.5 - 31 kg/meter square (m^2) (inclusive).
* Male or Female. Females A female participant is eligible to participate if she is not pregnant (as confirmed by a negative serum or urine human chorionic gonadotrophin (hCG) test), not lactating, and at least one of the following conditions applies: Non-reproductive potential defined as: Pre-menopausal females with one of the following: Documented tubal ligation or Documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral tubal occlusion or Hysterectomy or Documented Bilateral Oophorectomy; Postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the consent form and in the protocol.

Exclusion Criteria:

* ALT and bilirubin >1.5x upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent [%]).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Participants with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Participants with a history of cholecystectomy, peptic ulceration, inflammatory bowel disease or pancreatitis should be excluded.
* Corrected QT (QTc) interval according to Fridericia's formula (QTcF) > 450 milli-seconds (msec).

Notes:

1. The QTc is the QT interval corrected for heart rate according to Fridericia's formula, machine-read or manually over-read.
2. The specific formula that will be used to determine eligibility and discontinuation for an individual participant should be determined prior to initiation of the study. In other words, several different formulae cannot be used to calculate the QTc for an individual participant and then the lowest QTc value used to include or discontinue the participant from the trial.
3. For purposes of data analysis, Corrected QT interval according to Bazett's formula (QTcB), QTcF, another QT correction formula, or a composite of available values of QTc will be used as specified in the Reporting and Analysis Plan (RAP).

   * Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication until completion of the follow-up visit, unless in the opinion of the Investigator and Medical Monitor the medication will not interfere with the study procedures or compromise participant safety.
   * History of regular alcohol consumption within 6 months of the study defined as: An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 millilitre [mL]) of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
   * Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
   * Consumption of red wine, Seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medications.
   * History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
   * Creatinine clearance (CrCL) <60 mL/minutes (min).
   * Presence of hepatitis B surface antigen (HBsAg), positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study treatment.
   * A positive pre-study drug/alcohol screen.
   * A positive test for HIV antibody.
   * Where participation in the study would result in donation of blood or blood product in excess of 500 mL within 56 days.
   * The participant has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
   * Exposure to more than four new chemical entities within 12 months prior to the first dosing day.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01-01; Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States

REFERENCES:
- [Derived] Adkison K, Wolstenholme A, Lou Y, Zhang Z, Eld A, Perger T, Vangerow H, Hayward K, Shaefer M, McCoig C. Effect of Sorbitol on the Pharmacokinetic Profile of Lamivudine Oral Solution in Adults: An Open-Label, Randomized Study. Clin Pharmacol Ther. 2018 Mar;103(3):402-408. doi: 10.1002/cpt.943. Epub 2017 Dec 11. PMID 29150845

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Sixteen subjects were randomized to one of the 4 treatment sequences separated by >=7 day washout between doses.
Groups:
- Treatment Sequence 1: ADBC; Treatment Sequence 2: BACD; Treatment Sequence 3: CBDA; Treatment Sequence 4: DCAB: Participants were randomized to receive a single dose of each of the four treatments where A: Lamivudine 300 mg, B: Lamivudine 300 mg+ Sorbitol 3.2 g, C: Lamivudine 300 mg+ Sorbitol 10.2 g, D: Lamivudine 300 mg+ Sorbitol 13.4 g. All doses were administered after an overnight fast and there was >=7days washout between each period
Period: Overall Study
Arm/Group | Treatment Sequence 1: ADBC | Treatment Sequence 2: BACD | Treatment Sequence 3: CBDA | Treatment Sequence 4: DCAB
Started | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Treatment Groups Combined: Sixteen participants were randomized to receive one of the following 4 treatment sequences : Treatment sequence 1 : ABCD; Treatment sequence 2: DABC; Trearment sequence 3: BCDA; Treatment sequence 4: CDAB; where A: Lamivudine 300 mg, B: Lamivudine 300 mg+ Sorbitol 3.2 g, C: Lamivudine 300 mg+ Sorbitol 10.2 g, D: Lamivudine 300 mg+ Sorbitol 13.4 g.
Arm/Group | All Treatment Groups Combined
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (12.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  African American/African Heritage | 6
  White - White/Caucasian/European Heritage | 10

OUTCOME MEASURES:

1. Primary Outcome: Plasma Lamivudine Area Under the Plasma Concentration Time Curve (AUC) From Time Zero to the Last Quantifiable Time Point (AUC[0-t]), AUC From Time Zero Extrapolated to Infinity (AUC[0-inf]) and AUC From Time Zero to 24 Hours (AUC[0-24])
Description: Serial blood sample were collected at Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose in each treatment period. AUC was determined using the trapezoidal rule. Analysis of variance (ANOVA), considering treatment and period as fixed effects and participant as random effect, was performed using Mixed Linear Models procedure to compare the plasma lamivudine Pharmacokinetic (PK) parameters.
Time Frame: Day 1 to Day 3 in each treatment period
Population: PK Summary Population: defined as participants who had valid lamivudine PK parameter estimates from both reference and test treatments. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour (h)*microgram (mcg)/milliliter (mL)
Groups:
- A: Lamivudine 300 mg: After overnight fasting, participants received a single dose of treatment A: lamivudine 300 milligram (mg) (30 millilitre (mL) of 10 mg/mL oral solution) in one of the four treatment periods according to randomisation. There was a washout period of 7 days between the doses.
- B: Lamivudine 300 mg + Sorbitol 3.2 g: After overnight fasting, participants received a single dose of treatment B: lamivudine 300 mg (30 mL of 10 mg/mL oral solution) and an oral solution containing sorbitol 3.2 grams (g) in one of the four treatment periods according to randomisation. There was a washout period of 7 days between the doses.
- C: Lamivudine 300 mg + Sorbitol 10.2 g: After overnight fasting, participants received a single dose of treatment C: lamivudine 300 mg (30 mL of 10 mg/mL oral solution) and an oral solution containing sorbitol 10.2 g in one of the four treatment periods according to randomisation. There was a washout period of 7 days between the doses.
- D: Lamivudine 300 mg + Sorbitol 13.4 g: After overnight fasting, participants received a single dose of treatment D: lamivudine 300 mg (30 mL of 10 mg/mL oral solution) and an oral solution containing sorbitol 13.4 g in one of the four treatment periods according to randomisation. There was a washout period of 7 days between the doses.
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
hour (h)*microgram (mcg)/milliliter (mL)
  AUC (0-inf); n=16, 14, 16, 13 | 13.2 (22.3) | 11.3 (21.2) | 8.93 (22.1) | 8.60 (24.1)
  AUC (0-24) ; n=16, 16, 16, 16 | 12.4 (23.6) | 9.96 (22.6) | 7.54 (23.7) | 6.91 (28.9)
  AUC (0-t) ; n=16, 16, 16, 16 | 12.9 (23.0) | 10.6 (21.6) | 8.21 (22.9) | 7.55 (26.8)
Statistical Analysis 1: Comparison: A: Lamivudine 300 mg vs B: Lamivudine 300 mg + Sorbitol 3.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 0.855, 90% CI 2-sided [0.799 to 0.914] — AUC (0-inf) comparison
Statistical Analysis 2: Comparison: A: Lamivudine 300 mg vs C: Lamivudine 300 mg + Sorbitol 10.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 0.677, 90% CI 2-sided [0.635 to 0.721] — AUC (0-inf) comparision
Statistical Analysis 3: Comparison: A: Lamivudine 300 mg vs D: Lamivudine 300 mg + Sorbitol 13.4 g; Test type: Superiority or Other; ANCOVA; Ratio = 0.637, 90% CI 2-sided [0.594 to 0.682] — AUC (0-inf) comparision
Statistical Analysis 4: Comparison: A: Lamivudine 300 mg vs B: Lamivudine 300 mg + Sorbitol 3.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 0.803, 90% CI 2-sided [0.747 to 0.864] — AUC (0-24) comparision
Statistical Analysis 5: Comparison: A: Lamivudine 300 mg vs C: Lamivudine 300 mg + Sorbitol 10.2 g; Test type: Superiority or Other; ANOVA; Ratio = 0.608, 90% CI 2-sided [0.566 to 0.655] — AUC (0-24) comparision
Statistical Analysis 6: Comparison: A: Lamivudine 300 mg vs D: Lamivudine 300 mg + Sorbitol 13.4 g; Test type: Superiority or Other; ANCOVA; Ratio = 0.557, 90% CI 2-sided [0.518 to 0.599] — AUC (0-24) comparision
Statistical Analysis 7: Comparison: A: Lamivudine 300 mg vs B: Lamivudine 300 mg + Sorbitol 3.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 0.819, 90% CI 2-sided [0.766 to 0.876] — AUC (0-t) comparision
Statistical Analysis 8: Comparison: A: Lamivudine 300 mg vs C: Lamivudine 300 mg + Sorbitol 10.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 0.636, 90% CI 2-sided [0.595 to 0.680] — AUC (0-t) comparision
Statistical Analysis 9: Comparison: A: Lamivudine 300 mg vs D: Lamivudine 300 mg + Sorbitol 13.4 g; Test type: Superiority or Other; ANCOVA; Ratio = 0.585, 90% CI 2-sided [0.548 to 0.626] — AUC (0-t) comparision

2. Primary Outcome: Plasma Lamivudine Maximum Observed Concentration (Cmax), Concentration at 24 Hour (h) Post-dose (C24) and Last Measurable Concentration (Ct)
Description: Serial blood sample were collected at Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose in each treatment period. Time of the last measurable concentration (t) was 48 hours for all participants and all treatments. ANOVA, considering treatment and period as fixed effects and participant as random effect, was performed using Mixed Linear Models procedure to compare the plasma lamivudine PK parameters.
Time Frame: Day 1 to Day 3 in each treatment period
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
mcg/mL
  C24 | 0.036 (25.1) | 0.036 (31.1) | 0.041 (21.8) | 0.039 (21.6)
  Ct | 0.013 (28.4) | 0.017 (26.3) | 0.019 (38.7) | 0.018 (51.5)
  Cmax | 3.34 (34.9) | 2.42 (32.7) | 1.60 (27.2) | 1.52 (30.9)
Statistical Analysis 1: Comparison: A: Lamivudine 300 mg vs B: Lamivudine 300 mg + Sorbitol 3.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 0.993, 90% CI 2-sided [0.916 to 1.08] — C24 comparison
Statistical Analysis 2: Comparison: A: Lamivudine 300 mg vs C: Lamivudine 300 mg + Sorbitol 10.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 1.12, 90% CI 2-sided [1.03 to 1.21] — C24 comparision
Statistical Analysis 3: Comparison: A: Lamivudine 300 mg vs D: Lamivudine 300 mg + Sorbitol 13.4 g; Test type: Superiority or Other; ANCOVA; Ratio = 1.09, 90% CI 2-sided [1.000 to 1.18] — C24 comparision
Statistical Analysis 4: Comparison: A: Lamivudine 300 mg vs B: Lamivudine 300 mg + Sorbitol 3.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 1.33, 90% CI 2-sided [1.13 to 1.56] — Ct comparision
Statistical Analysis 5: Comparison: A: Lamivudine 300 mg vs C: Lamivudine 300 mg + Sorbitol 10.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 1.46, 90% CI 2-sided [1.25 to 1.71] — Ct comparision
Statistical Analysis 6: Comparison: A: Lamivudine 300 mg vs D: Lamivudine 300 mg + Sorbitol 13.4 g; Test type: Superiority or Other; ANCOVA; Ratio = 1.39, 90% CI 2-sided [1.18 to 1.63] — Ct comparision
Statistical Analysis 7: Comparison: A: Lamivudine 300 mg vs B: Lamivudine 300 mg + Sorbitol 3.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 0.724, 90% CI 2-sided [0.657 to 0.798] — Cmax comparision
Statistical Analysis 8: Comparison: A: Lamivudine 300 mg vs C: Lamivudine 300 mg + Sorbitol 10.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 0.479, 90% CI 2-sided [0.434 to 0.527] — Cmax comparision
Statistical Analysis 9: Comparison: A: Lamivudine 300 mg vs D: Lamivudine 300 mg + Sorbitol 13.4 g; Test type: Superiority or Other; ANCOVA; Ratio = 0.454, 90% CI 2-sided [0.412 to 0.500] — Cmax comparision

3. Primary Outcome: Lamivudine Elimination Half-life in Plasma (t1/2)
Description: Serial blood sample were collected at Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose in each treatment period. ANOVA, considering treatment and period as fixed effects and participant as random effect, was performed using Mixed Linear Models procedure to compare the plasma lamivudine t1/2.
Time Frame: Day 1 to Day 3 in each treatment period
Population: PK Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour (Hr)
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 14 | 16 | 13
Hour (Hr) | 13.9 (20.9) | 19.0 (40.6) | 21.2 (47.3) | 17.3 (48.6)
Statistical Analysis 1: Comparison: A: Lamivudine 300 mg vs B: Lamivudine 300 mg + Sorbitol 3.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 1.37, 90% CI 2-sided [1.11 to 1.69]
Statistical Analysis 2: Comparison: A: Lamivudine 300 mg vs C: Lamivudine 300 mg + Sorbitol 10.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 1.53, 90% CI 2-sided [1.25 to 1.88]
Statistical Analysis 3: Comparison: A: Lamivudine 300 mg vs D: Lamivudine 300 mg + Sorbitol 13.4 g; Test type: Superiority or Other; ANCOVA; Ratio = 1.29, 90% CI 2-sided [1.04 to 1.61]

4. Primary Outcome: Plasma Lamivudine Apparent Oral Clearance (CL/F)
Description: Serial blood sample were collected at Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose in each treatment period. ANOVA, considering treatment and period as fixed effects and participant as random effect, was performed using Mixed Linear Models procedure to compare the plasma lamivudine CL/F
Time Frame: Day 1 to Day 3 in each treatment period
Population: PK Summary Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)/hr
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 14 | 16 | 13
Liter (L)/hr | 22.738 (22.3) | 26.621 (21.2) | 33.608 (22.1) | 34.875 (24.1)
Statistical Analysis 1: Comparison: A: Lamivudine 300 mg vs B: Lamivudine 300 mg + Sorbitol 3.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 1.170, 90% CI 2-sided [1.094 to 1.251]
Statistical Analysis 2: Comparison: A: Lamivudine 300 mg vs C: Lamivudine 300 mg + Sorbitol 10.2 g; Test type: Superiority or Other; ANCOVA; Ratio = 1.478, 90% CI 2-sided [1.386 to 1.576]
Statistical Analysis 3: Comparison: A: Lamivudine 300 mg vs D: Lamivudine 300 mg + Sorbitol 13.4 g; Test type: Superiority or Other; ANCOVA; Ratio = 1.571, 90% CI 2-sided [1.466 to 1.684]

5. Primary Outcome: Time to Observed Maximum Lamivudine Plasma Concentration (Tmax), Time of Last Measurable Plasma Concentration (Tlast) and Absorption Lag Time in Plasma (Tlag)
Description: Serial blood sample were collected at Pre-dose; 0.25, 0.5, 0.75, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, 24, 36 and 48 hours post-dose in each treatment period.
Time Frame: Day 1 to Day 3 in each treatment period
Measure: Median (Full Range); unit: Hr
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
Hr
  tmax | 0.75 [0.50 to 1.50] | 1.000 [0.50 to 1.50] | 1.00 [0.50 to 2.50] | 1.26 [0.50 to 3.00]
  tlast | 48.00 [48.00 to 48.22] | 48.00 [47.50 to 48.08] | 48.00 [47.57 to 48.03] | 48.00 [48.00 to 48.07]
  tlag | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00] | 0.000 [0.00 to 0.00]

6. Secondary Outcome: Number of Participants With Any Adverse Events (AEs) and Any Serious Adverse Events (SAE)
Description: An AE is any untoward medical occurrence, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that at any dose results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect or event that may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in the above definition.
Time Frame: Up to 5 Weeks
Population: Safety Population: defined as all participants who enrolled into the study and received at least one dose of study drug.
Measure: Number; unit: Participants
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
Participants
  AEs | 1 | 2 | 1 | 1
  SAEs | 0 | 0 | 0 | 0

7. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Change from Baseline for pulse rate was calculated as the post-dose visit value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/period.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population.Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: Beats/min
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
Beats/min
  Day 3; n=15, 16, 16, 16 | 6.5 (3.42) | 3.9 (14.3) | 6.0 (6.86) | 7.4 (8.57)
  Follow up; n=16, 16, 16, 16 | 5.8 (6.41) | 5.8 (6.41) | 5.8 (6.41) | 5.8 (6.41)

8. Secondary Outcome: Change From Baseline in Body Temperature
Description: Change from Baseline for body temperature was calculated as the post-dose visit value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/period.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Degree centigrade
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
Degree centigrade
  Day 3 | 0.03 (0.252) | 0.07 (0.189) | 0.08 (0.183) | -0.03 (0.145)
  Follow up | -0.01 (0.365) | -0.01 (0.365) | -0.01 (0.365) | -0.01 (0.365)

9. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Change from Baseline for DBP and SBP was calculated as the post-dose visit value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/period.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population. Only those participants available at the specified time points were analyzed (represented by n=X, X in the category titles).
Measure: Mean (Standard Deviation); unit: millimeter of mercury (mmHg)
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
millimeter of mercury (mmHg)
  DBP, Day 3; n=15, 16, 16, 16 | 5.1 (6.41) | 4.5 (4.13) | 2.1 (7.46) | 5.6 (4.87)
  DBP, Follow up; n=16, 16, 16, 16 | 4.6 (6.54) | 4.6 (6.54) | 4.6 (6.54) | 4.6 (6.54)
  SBP, Day 3; n=15, 16, 16, 16 | 3.6 (9.84) | 3.1 (8.01) | 5.1 (7.19) | 5.3 (7.38)
  SBP, Follow up; n=16, 16, 16, 16 | 7.4 (7.78) | 7.4 (7.78) | 7.4 (7.78) | 7.4 (7.78)

10. Secondary Outcome: Number of Participants With Treatment Emergent Laboratory Abnormality Grade
Description: Division of Acquired immune deficiency syndrome (DAIDS) Table AE grades 1, 2, 3, and 4 of laboratory abnormalities were applied and grade were summarized by treatment and day and were listed by participant, treatment, day, and actual date and time. Treatment emergent grades are defined as any new toxicity grades or the worsened grades compared to Baseline grade. Treatment emergent lab abnormality Grade 1 for aspartate aminotransferase and sodium at follow-up visit are summarized.
Time Frame: Up to Week 5
Population: Safety Population
Measure: Number; unit: Participants
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
Participants
  Aspartate Aminotransferase | 1 | 1 | 1 | 1
  Sodium | 1 | 1 | 1 | 1

11. Secondary Outcome: Change From Baseline in Erythrocytes
Description: Blood samples were collected at Day -1, Day 3 of every treatment period and at follow-up. Change from Baseline for erythrocytes was calculated as the post-dose visit value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/Period. Day -1 presented the Baseline absolute values; Day 3 and Follow-Up presented the changes from Baseline.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
10^12 cells/L
  Day 3 | 0.351 (0.298) | 0.389 (0.200) | 0.339 (0.257) | 0.380 (0.243)
  Follow up | 0.142 (0.148) | 0.142 (0.148) | 0.142 (0.148) | 0.142 (0.148)

12. Secondary Outcome: Change From Baseline in Hematocrit
Description: Blood samples were collected at Day -1, Day 3 of every treatment period and at follow-up. Change from Baseline for hematocrit was calculated as the post-dose visit value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/period. Day -1 presented the Baseline absolute values; Day 3 and Follow-Up presented the changes from Baseline.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Fraction of 1
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
Fraction of 1
  Day 3 | 0.0338 (0.02429) | 0.0378 (0.02206) | 0.0308 (0.01993) | 0.0353 (0.01892)
  Follow up | 0.0091 (0.01254) | 0.0091 (0.01254) | 0.0091 (0.01254) | 0.0091 (0.01254)

13. Secondary Outcome: Change From Baseline in Hemoglobin
Description: Blood samples were collected at Day -1, Day 3 of every treatment period and at follow-up. Change from Baseline for hemoglobin was calculated as the post-dose visit value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/period. Day -1 presented the Baseline absolute values; Day 3 and Follow-Up presented the changes from Baseline.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: G/L
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
G/L
  Day 3 | 10.1 (8.05) | 10.9 (5.26) | 9.8 (6.44) | 9.9 (5.83)
  Follow up | 3.4 (4.57) | 3.4 (4.57) | 3.4 (4.57) | 3.4 (4.57)

14. Secondary Outcome: Change From Baseline in Mean Corpuscular Hemoglobin (MCH)
Description: Blood samples were collected at Day -1, Day 3 of every treatment period and at follow-up. Change from Baseline for MCH was calculated as the post-dose visit value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/period. Day -1 presented the Baseline absolute values; Day 3 and Follow-Up presented the changes from Baseline.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
Picogram
  Day 3 | 0.02 (0.500) | -0.03 (0.419) | 0.06 (0.403) | -0.24 (0.622)
  Follow up | -0.14 (0.567) | -0.14 (0.567) | -0.14 (0.567) | -0.14 (0.567)

15. Secondary Outcome: Change From Baseline in Mean Corpuscular Volume (MCV)
Description: Blood samples were collected at Day -1, Day 3 of every treatment period and at follow-up. Change from Baseline for MCV was calculated as the post-dose visit value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/period. Day -1 presented the Baseline absolute values; Day 3 and Follow-Up presented the changes from Baseline.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Femtoliter
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
Femtoliter
  Day 3 | 0.71 (1.95) | 0.63 (1.89) | 0.35 (2.06) | 0.44 (1.54)
  Follow up | -0.77 (1.55) | -0.77 (1.55) | -0.77 (1.55) | -0.77 (1.55)

16. Secondary Outcome: Change From Baseline in Platelets, Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils
Description: Blood samples were collected at Day -1, Day 3 of every treatment period and at follow-up. Change from Baseline for platelets, neutrophils, lymphocytes, monocytes, eosinophils, basophils were calculated as the post-dose visit value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/period. Day -1 presented the Baseline absolute values; Day 3 and Follow-Up presented the changes from Baseline.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
10^9 cells/L
  Platelets, Day 3 | 19.2 (20.69) | 13.9 (15.75) | 13.8 (20.92) | 6.1 (24.65)
  Platelets, Follow up | 2.3 (19.36) | 2.3 (19.36) | 2.3 (19.36) | 2.3 (19.36)
  Neutrophils, Day 3 | 0.35 (0.612) | 0.42 (0.733) | 0.53 (0.603) | 0.31 (0.979)
  Neutrophils, Follow up | -0.12 (0.717) | -0.12 (0.717) | -0.12 (0.717) | -0.12 (0.717)
  Lymphocytes, Day 3 | 0.10 (0.432) | 0.17 (0.338) | 0.00 (0.446) | -0.03 (0.466)
  Lymphocytes, Follow up | -0.08 (0.371) | -0.08 (0.371) | -0.08 (0.371) | -0.08 (0.371)
  Monocytes, Day 3 | 0.01 (0.085) | 0.03 (0.060) | -0.02 (0.122) | -0.01 (0.112)
  Monocytes, Follow up | -0.08 (0.134) | -0.08 (0.134) | -0.08 (0.134) | -0.08 (0.134)
  Eosinophils, Day 3 | -0.03 (0.070) | -0.02 (0.075) | -0.04 (0.062) | -0.03 (0.070)
  Eosinophils, Follow up | -0.01 (0.068) | -0.01 (0.068) | -0.01 (0.068) | -0.01 (0.068)
  Basophils, Day 3 | -0.01 (0.025) | 0.00 (0.000) | -0.01 (0.025) | 0.00 (0.037)
  Basophils, Follow up | -0.01 (0.025) | -0.01 (0.025) | -0.01 (0.025) | -0.01 (0.025)

17. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen (BUN), Sodium, Potassium, Glucose, Calcium
Description: Blood samples were collected at Day -1, Day 3 of every treatment period and at follow-up. Change from Baseline for BUN, sodium, potassium, glucose, calcium were calculated as the post-dose visit value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/period. Day -1 presented the Baseline absolute values; Day 3 and Follow-Up presented the changes from Baseline.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: millimole (mmol)/L
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
millimole (mmol)/L
  BUN, Day 3 | -0.0892 (1.08675) | -0.5578 (0.93974) | 0.0223 (1.05476) | 0.0446 (1.38496)
  BUN, Follow up | -0.4909 (1.00870) | -0.4909 (1.00870) | -0.4909 (1.00870) | -0.4909 (1.00870)
  Sodium, Day 3 | -2.4 (1.71) | -1.2 (1.42) | -2.6 (1.59) | -2.0 (1.63)
  Sodium, Follow up | -0.1 (2.03) | -0.1 (2.03) | -0.1 (2.03) | -0.1 (2.03)
  Potassium, Day 3 | 0.06 (0.418) | 0.09 (0.481) | 0.19 (0.382) | 0.06 (0.386)
  Potassium, Follow up | 0.02 (0.387) | 0.02 (0.387) | 0.02 (0.387) | 0.02 (0.387)
  Glucose, Day 3 | -0.05897 (0.496601) | 0.05550 (0.342125) | 0.01388 (0.342425) | -0.03122 (0.657300)
  Glucose, Follow up | 0.33994 (0.546377) | 0.33994 (0.546377) | 0.33994 (0.546377) | 0.33994 (0.546377)
  Calcium Day 3 | 0.0906 (0.11614) | 0.1141 (0.08214) | 0.1141 (0.07744) | 0.0875 (0.07583)
  Calcium, Follow up | 0.0328 (0.05379) | 0.0328 (0.05379) | 0.0328 (0.05379) | 0.0328 (0.05379)

18. Secondary Outcome: Change From Baseline in Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) and Alkaline Phosphates
Description: Blood samples were collected at Day -1, Day 3 of every treatment period and at follow-up. Change from Baseline for AST, ALT and alkaline phosphatase were calculated as the post-dose visit value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/period. Day -1 presented the Baseline absolute values; Day 3 and Follow-Up presented the changes from Baseline.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Unit (U)/L
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
Unit (U)/L
  AST, Day 3 | -3.1 (4.84) | -3.5 (3.67) | -2.3 (2.44) | -19.1 (68.13)
  AST, Follow up | 1.1 (15.86) | 1.1 (15.86) | 1.1 (15.86) | 1.1 (15.86)
  ALT, Day 3 | -2.2 (5.78) | -2.7 (4.16) | -2.2 (2.59) | -2.5 (7.05)
  ALT, Follow up | 0.4 (8.97) | 0.4 (8.97) | 0.4 (8.97) | 0.4 (8.97)
  Alkaline phosphatatse, Day 3 | -0.4 (7.96) | 1.1 (6.24) | 1.5 (8.45) | -0.2 (7.37)
  Alkaline phosphatase, Follow up | 1.2 (7.01) | 1.2 (7.01) | 1.2 (7.01) | 1.2 (7.01)

19. Secondary Outcome: Change From Baseline in Creatinine, Total Bilirubin and Direct Bilirubin
Description: Blood samples were collected at Day -1, Day 3 of every treatment period and at follow-up. Change from Baseline for creatinine and direct bilirubin were calculated as the post-dose visit value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/period. Change from Baseline in total bilirubine was not assessed. Day -1 presented the Baseline absolute values; Day 3 and Follow-Up presented the changes from Baseline.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: micromole (umol)/L
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
micromole (umol)/L
  Creatinine, Day 3 | 3.86759 (9.112270) | 2.21005 (6.847589) | 4.42010 (7.217993) | 0.55251 (6.011986)
  Creatinine, Follow up | 0.00000 (7.217993) | 0.00000 (7.217993) | 0.00000 (7.217993) | 0.00000 (7.217993)
  Direct bilirubin, Day 3 | 0.641 (0.8550) | 0.107 (1.3200) | 0.107 (0.7567) | 0.321 (1.1202)
  Direct bilirubin, Follow up | 0.107 (1.4602) | 0.107 (1.4602) | 0.107 (1.4602) | 0.107 (1.4602)

20. Secondary Outcome: Change From Baseline in Albumin
Description: Blood samples were collected at Day -1, Day 3 of every treatment period and at follow-up. Change from Baseline for albumin was calculated as the post-dose Visit Value minus the value at Baseline, at Day 3 and Follow-up. Baseline value used in the analysis was the latest pre-dose values on Day 1 of each treatment/Period. Day -1 presented the Baseline absolute values; Day 3 and Follow-Up presented the changes from Baseline.
Time Frame: Baseline and up to 5 weeks
Population: Safety Population
Measure: Mean (Standard Deviation); unit: G//L
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Number analyzed (Participants) | 16 | 16 | 16 | 16
G//L
  Day 3 | 1.8 (2.43) | 2.3 (1.58) | 2.1 (2.38) | 2.1 (2.09)
  Follow up | 0.6 (1.63) | 0.6 (1.63) | 0.6 (1.63) | 0.6 (1.63)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study medication until follow-up (up to 5 weeks).
Description: On-treatment SAEs and non-serious AEs are reported for Safety Population.
Arm/Group | A: Lamivudine 300 mg | B: Lamivudine 300 mg + Sorbitol 3.2 g | C: Lamivudine 300 mg + Sorbitol 10.2 g | D: Lamivudine 300 mg + Sorbitol 13.4 g
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 1/16 | 2/16 | 1/16 | 1/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A: Lamivudine 300 mg (N=16) | B: Lamivudine 300 mg + Sorbitol 3.2 g (N=16) | C: Lamivudine 300 mg + Sorbitol 10.2 g (N=16) | D: Lamivudine 300 mg + Sorbitol 13.4 g (N=16)
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.